CLINICAL TRIAL: NCT07358871
Title: Testing the Effects of Music on Short-Term Changes in Affective Valence, Arousal, and RPE, Long Term Changes in Enjoyment, Motivation, and Commitment to Physical Activity, and Step Counts in Children
Brief Title: Testing the Effects of Music on Short and Long Term Psychological Outcomes and Step Counts in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Kyle A. Kercher, Assistant Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 27934
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Music Exposure
Keywords: Sport Based Youth Development; Children; Asynchronous Music

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Music (Active Comparator): The control group will participate in the Hoosier Sport program during their school's physical education class, which consists of sport curriculums, leadership development, and health lessons. Participants will complete this with no exposure to music.
  Interventions: Behavioral: No Music Exposure
- Music (Experimental): The experimental group will participate in the Hoosier Sport program during their school's physical education class, which consists of sport curriculums, leadership development, and health lessons. This group will complete this program with asynchronous music during drills and games.
  Interventions: Behavioral: Music in Sport Based Youth Development

INTERVENTIONS:
Behavioral: Music in Sport Based Youth Development — The intervention being tested is the use of music during Hoosier Sport lessons. Asynchronous music that is 120+ beats per minute, generally upbeat, and school appropriate will be played during the experimental group's drills and games. The experimental group will be exposed to this music for each lesson throughout the 8-week intervention.
  Arms: Music
Behavioral: No Music Exposure — This group will participate in the Hoosier Sport program with no exposure to music.
  Arms: No Music

SUMMARY:
The goal of this clinical trial is to investigate whether asynchronous music can improve outcomes of an 8-week long sport based youth development program. The main questions it aims to answer are:

* Does music increase step count during each lesson?
* Does music create a larger improvement in affective valence, arousal, and rate of perceived exertion (RPE) during each lesson?
* Does music create a long term improvement in enjoyment, commitment, and intrinsic motivation to exercise?
* Does music show more improvement among sedentary participants versus active participants? Researchers will compare the results from the experimental group, which is exposed to music, to the control group, which is not exposed to music.

Participants will:

* Participate in the sport based youth development program, Hoosier Sport, during their school's physical education class once a week for 8 weeks.
* Respond to 3 questions regarding affective valence, arousal, and RPE before and after each lesson.
* Complete a detailed survey regarding basic demographics, their music preferences, enjoyment of exercise, motivation to exercise, commitment to exercise, and current activity levels before the intervention.
* Complete the same sections regarding enjoyment of exercise, motivation to exercise, and commitment to exercise at a mid and end point of the intervention.

DETAILED DESCRIPTION:
30+ students (5th-6th grade) from Clear Creek Christian School (CCCS) will be recruited to participate in the present study for the Spring of 2026. This group will participate in Hoosier Sport lessons that take place during their scheduled PE time at CCCS once a week for 8 weeks.

Hoosier Sport intervention components include sport participation and leadership development activities. Hoosier Sport is a part of Clear Creek Christian School's regular PE classes and is separate from this study procedure. Classes will be divided into classes with music (experimental group) and classes without music (control group) and will remain in these categories for the duration of the intervention. Students will be blinded to the purpose of this experiment to avoid performance bias and the expectation of music during classes in the control group. The Hoosier Sport curriculum will remain the same for both groups. In the classes with music, music will be played during drills and games and paused during instruction. The music will be upbeat, 120+ beats per minute, and school appropriate. The research team will incorporate students' music preferences where possible.

Once participants express interest in joining the study, the research team will set up a phone call to obtain consent and assent. There will be a survey for participants to take prior to the start of the intervention. Included in this survey are questions about basic demographics, music preferences, the physical activity section of the Global School Based Health Survey (GSHS) to determine active versus sedentary students, the Physical Activity Enjoyment Scale Short Version (PACES-S) to determine their enjoyment of physical activity, the enjoyment/interest subsection of the Intrinsic Motivation Inventory (IMI) to determine levels of motivation to exercise, and the Commitment to Physical Activity Scale for Adolescents (CPASA) to determine commitment to exercise. Before and after each Hoosier Sport lesson, the children will complete the Feeling Scale, Felt Arousal Scale, and rate of perceived exertion (1 question each) to determine their current affect, activation levels, and effort. The students will complete the PACES-S, IMI Enjoyment/Interest subsection, and CPASA after week 4 and week 8 of the intervention. During each lesson, students will wear Yamax SW-200 pedometers to track their step counts, which will be returned at the end of each lesson.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in 5th or 6th grade at Clear Creek Elementary
* have parental consent to participate
* agree to study participation (verbal assent)
* planning to attend all school days during the 8-week program period
* enrolled in PE for the semester

Exclusion Criteria:

* not already participating in Hoosier Sport/PE at Clear Creek Christian School

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Step Count | 8 weeks
  Step counts during Hoosier Sport lessons will be measured using Yamax SW-200 Digi Walker pedometers.

SECONDARY OUTCOMES:
Affective Valence | 8 weeks
  Participants will complete the Feeling Scale before and after each Hoosier Sport lesson to measure any changes in affective valence.
Activation | 8 weeks
  Participants will complete the Felt Arousal Scale before and after each Hoosier Sport lesson to measure any changes in their activation during each session.
Rate of Perceived Exertion | 8 weeks
  Participants will specify their rate of perceived exertion after each Hoosier Sport lesson to determine their effort during the session.
Commitment to Physical Activity | 8 weeks
  Participants will fill out the Commitment to Physical Activity Scale for Adolescents pre, mid, and post intervention to determine their commitment to physical activity.
Enjoyment of Physical Activity | 8 weeks
  Participants will complete the Physical Activity Enjoyment Scale Short Version pre, mid, and post intervention to determine how much they enjoy physical activity.
Motivation to Exercise | 8 weeks
  Participants will complete the Intrinsic Motivation Inventory- Enjoyment/Interest Subsection pre, mid, and post intervention to determine their levels of motivation to exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- Clear Creek Christian School, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robbins LB, Ling J, Wesolek SM, Kazanis AS, Bourne KA, Resnicow K. Reliability and Validity of the Commitment to Physical Activity Scale for Adolescents. Am J Health Promot. 2017 Jul;31(4):343-352. doi: 10.4278/ajhp.150114-QUAN-665. Epub 2016 Nov 17. PMID 26730556
- [Background] Chen C, Weyland S, Fritsch J, Woll A, Niessner C, Burchartz A, Schmidt SCE, Jekauc D. A Short Version of the Physical Activity Enjoyment Scale: Development and Psychometric Properties. Int J Environ Res Public Health. 2021 Oct 20;18(21):11035. doi: 10.3390/ijerph182111035. PMID 34769552
- [Background] Bastos V, Rodrigues F, Davis P, Teixeira DS. Assessing affective valence and activation in resistance training with the feeling scale and the felt arousal scale: A systematic review. PLoS One. 2023 Nov 16;18(11):e0294529. doi: 10.1371/journal.pone.0294529. eCollection 2023. PMID 37972201
- [Background] Terry PC, Karageorghis CI, Curran ML, Martin OV, Parsons-Smith RL. Effects of music in exercise and sport: A meta-analytic review. Psychol Bull. 2020 Feb;146(2):91-117. doi: 10.1037/bul0000216. Epub 2019 Dec 5. PMID 31804098
- [Background] Barney, D., & Prusak, K. A. (2015). Effects of music on physical activity rates of elementary physical education students. The Physical Educator, 72, 236-244.
- [Background] Bassett, J., West, S., & Shores, K. (2011). The Effects of Asynchronous Music on the Physical Activities of Youth in Supervised Recreation Activities. Journal of Park & Recreation Administration, 29(1).